CLINICAL TRIAL: NCT03336788
Title: Virtual Reality Combined With rTMS for the Treatment of Depression : a Randomized Clinical Trial.
Acronym: TMS VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-21; 2016-A01115-46 (Registry Identifier: ID RCB)
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: the Treatment of Depression
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMS (Placebo Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS - ) MagPro®
- TMS with virtual reali (Active Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS - ) MagPro®; Device: virtual reality for displaying interactive virtual environments

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS - ) MagPro® — 20 sessions navigated with Conventional Transcranial Magnetic Stimulation
Device: virtual reality for displaying interactive virtual environments — 20 sessions navigated with virtual reality
  Arms: TMS with virtual reali

SUMMARY:
Depression is a mood disorder affecting an individual in its entirety, altering its emotional and intellectual functioning . The major form of depression is the most common psychiatric disorder in Western countries. It is considered to be the most expensive psychiatric neurological disease in Europe and is currently treated by different methods.

However, almost a third of depressed patients shows no clinical improvement. Advances in neuroscience and understanding of neuromodulation have enabled the emergence of new treatments such as the repetitive transcranial magnetic stimulation (rTMS) . It consists of modulating the neuronal activity of a targeted brain region through a magnetic field applied by a coil. Even though this form of treatment has proven to be effective, it appears that more than half of depressed patients exhibited little to no response to it.

As brain regions targeted by TMS may also be stimulated beforehand by sensory afferent signals, it was hypothesized that optimizing the effects of TMS with virtual reality is possible through the activation of these brain regions with sensory stimuli holding emotional valence (images, sounds) while using TMS concomitantly. Based on this new research premise, the investigators propose, in the context of an open and controlled clinical trial, to use a new media entitled virtual reality for displaying interactive virtual environments with positive emotional valence ( field of flowers, green valley) to a group of depressed patients undergoing TMS at the same time.

The study will include 66 depressed patients randomly assigned into two groups : TMS and Virtual Reality Versus TMS alone. Any differences in therapeutic efficacy between the two groups will be measured by questionnaires and brain functional imagery. This innovative and therapeutic approach will allow us to better understand the appropriate processes for modulating the neuronal activity in specific brain areas for treatment purposes.

ELIGIBILITY:
Inclusion Criteria:

* Criteria of resistant depression
* Age from 18 to 65 years old included.
* Primary diagnosis of major depression in subjects according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria.
* Informed consent and signed to participate in the study

Exclusion Criteria:

* Pregnant woman, parturient and nursing mothers.
* Absence of DSM-5 criteria for depression in subjects.
* Refusal to participate in the study.
* Modification of drug treatment in the month preceding inclusion.
* History of neurological pathology, head trauma or mental retardation.
* Presence of an addictive comorbidity.
* Presence of a major organic pathological.
* Presence of a contra-indication to virtual reality
* Presence of intracerebral ferro-metallic material, cochlear implant, pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-11-09 (Actual); Primary Completion 2019-11-09 (Estimated); Study Completion 2019-11-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the depression score in Montgomery-asberg Depression Rating Scale (MADRS). | 36 months
  a heteroevaluation scale of depressive semiology in 10 items. A decrease of at least 50% in initial score at the Montgomery-asberg Depression Rating Scale.

SECONDARY OUTCOMES:
Evaluation of The State Trait Anxiety Inventory Self-Questionnaire | 36 months
  40 items with, for each, 4 modalities of response, corresponding to degrees of intensity or frequency of the habitual or general emotional state of the patient. The calculated score varies between 20 and 80, a high score indicating the presence of anxiety. Anxiety will be assessed before the program begins and at the end of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Raphaëlle RICHIERI, PH, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France